CLINICAL TRIAL: NCT03618654
Title: Window of Opportunity for Durvalumab (MEDI4736) Plus Metformin Trial of in Squamous Cell Carcinoma of the Head and Neck
Brief Title: Durvalumab With or Without Metformin in Treating Participants With Head and Neck Squamous Cell Carcinoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18P.389; JT 12752 (Other: JeffTrial Number)
Record Dates: First submitted 2018-08-01; First posted 2018-08-07 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Oral Cavity Squamous Cell Carcinoma; Oropharyngeal Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Metformin; durvalumab; Immunoglobulin G

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A (durvalumab, metformin) (Experimental): Patients will take Metformin 500mg/day for 3 days. From day 4, 500mg twice daily and then in 3 days (day 7) dose escalation to 1000mg twice daily will be achieved. This will be taken until the day before surgery after dinner.
  Patients will receive 1500mg durvalumab (MEDI4736) via IV infusion
  Interventions: Drug: Metformin; Biological: Durvalumab
- Arm B (durvalumab) (Experimental): Patients will receive 1500mg durvalumab (MEDI4736) via IV infusion. Participants receive durvalumab as in Arm A in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Durvalumab

INTERVENTIONS:
Drug: Metformin — Given PO
  Other Names: 1,1-Dimethylbiguanide; 657-24-9; N,N-Dimethylimidodicarbonimidic Diamide
  Arms: Arm A (durvalumab, metformin)
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Kappa-chain; Human Monoclonal MEDI4736 Heavy Chain; MEDI4736; Immunoglobulin G1

SUMMARY:
This pilot phase I trial studies how well durvalumab given with or without metformin works in treating participants with head and neck squamous cell carcinoma. Monoclonal antibodies, such as durvalumab, may interfere with the ability of tumor cells to grow and spread. Metformin, a drug typically used for the treatment of diabetes, may help to reduce the metabolic activity of cancer cells and of surrounding supportive tissues. It is not yet known whether giving durvalumab with or without metformin may work better in treating participants with head and neck squamous carcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To investigate the combined effect of metformin and durvalumab on the immune tumor microenvironment, specifically with respect to alterations in T cell polarization (Th1/Th2 ratio) and tumor associated macrophage (TAM) (M1/M2 ratio) as measured by cytokine shifts in tumor specimens and peripheral blood.

SECONDARY OBJECTIVES:

I. To investigate the combined effect of metformin and durvalumab on the metabolic microenvironment, specifically with respect to alterations in immunohistochemical markers of the reverse Warburg effect.

II. To further characterize the alterations in intratumoral immune cell populations (effector T cells [Teff], regulatory T cells [Tregs], tumor associated macrophages [TAMs], and myeloid-derived suppressor cells [MDSC]).

III. To assess changes of the intratumoral immunophenotype and metabolism after exposure to durvalumab and metformin by transcriptome analysis using a ribonucleic acid-sequencing (RNA-seq) transcriptome analysis.

IV. To assess the efficacy of combined durvalumab and metformin treatment prior to surgery as determined by radiographic response and immune-related response criteria (irRC).

V. To assess the safety and tolerability of the combination of metformin and durvalumab.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed head and neck squamous cell carcinoma (HNSCC), with measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Any stage HNSCC of the 1) oral cavity, 2) oropharynx, 3) larynx, 4) hypopharynx, 5) nasal cavity/paranasal sinuses, 6) unknown primary, 7) skin considered to have resectable disease. Patients with recurrent disease that is amenable to surgery are eligible
* Performance status 0-1
* Must have a life expectancy of at least 12 weeks as judged by the treating physician
* Body weight >30 kg
* Absolute neutrophil count 1500/ul or more
* Platelets 100,000/ul or more
* Hemoglobin 9 g/dl or more
* Bilirubin less than or equal to 1.5 x the upper limit of normal (except subjects with Gilbert syndrome, who can have total bilirubin <3 mg/dl)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 2.5 x the upper limit of normal
* Glomerular filtration rate (GFR) greater than or equal to 40 ml/min using the Cockcroft-Gault formula or measured creatinine clearance using 24 hours urine collection
* Women of reproductive potential should have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]), which must also be confirmed as negative within 28 days of the start of study drugs
* Women of reproductive potential must use highly effective contraception methods to avoid pregnancy for 90 days after the last dose of study drugs. "Women of reproductive potential" is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes. In addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level less than 40 mIU/mL
* Men of reproductive potential who are sexually active with women of reproductive potential must use any contraceptive method with a failure rate of less than 1% per year. Men who are receiving the study medications will be instructed to adhere to contraception for 90 days after the last dose of study drugs. Men who are azoospermic do not require contraception
* Informed consent: All subjects must be able to comprehend and sign a written informed consent document

Exclusion Criteria:

* Patients with nasopharyngeal carcinoma or salivary gland primaries
* Any history of a sever hypersensitivity reaction to any monoclonal antibody
* Any history of allergy to the study drug components
* Any prior history of exposure to an anti PD-L1including durvalumab or PD1-directed therapy
* Patients who are already taking metformin, or who have taken metformin in the preceding 4 weeks
* Diabetic patients who are managed by taking metformin or insulin
* Major surgical procedure (as defined by the investigator) within 28 days prior to the first dose of durvalumab

  * Note: Local surgery of isolated lesions for palliative intent and biopsy procedures are acceptable
* Subjects who are on medication that are contraindicated with metformin under current Food and Drug Administration (FDA) recommendations; current recommendations reflect caution when metformin is used with insulin, sulfonylureas, and iodinated contrast dye
* Subjects who have received iodinated contrast dye less than 12 hours prior to screening meet a temporary exclusion criterion to receive metformin. These patients cannot start investigational metformin until 12 hours have elapsed from contrast administration. Subjects who are scheduled for iodinated contrast dye are not excluded but will be asked to hold their doses prior to dye administration
* Mean QT interval corrected for heart rate (QTc) greater than or equal to 470 ms calculated from 3 electrocardiograms (EKGs) using Fridericia's Correction
* Any concurrent malignancies; exceptions include- basal cell carcinoma of the skin, squamous cell carcinoma of the skin of a secondary location, superficial bladder cancer or in situ cervical cancer that has undergone potentially curative therapy. Patients with a history of other prior malignancy must have been treated with curative intent and must have remained disease-free for 2 years post-diagnosis
* Any unresolved toxicity National Cancer Institute NCI Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0 grade >= 2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria. Patients with grade >= 2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the study physician
* Any diagnosis of immunodeficiency or receiving systemic steroid therapy with a dose of >10 mg prednisone per day or equivalent or any other form of immunosuppressive therapy within 14 days of initiation of therapy, or a prior history of allogenic organ transplantation
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia
  * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
  * Patients with celiac disease controlled by diet alone
* Patients must not be receiving any other investigational agents
* Receipt of a live attenuated vaccine within 30 days prior to the first dose of drug on trial
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring adverse events (AEs) or compromise the ability of the patient to give written informed consent
* Patients must not be pregnant or breastfeeding
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis [TB] testing in line with local practice), hepatitis B virus (HBV) (known positive HBV surface antigen [HBsAg] result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
Immune cell polarization (Th1/Th2; M1/M2) | Up to 6 months
  The biomarker data will be compared for differences in means (or geometric means) between treatment arms using Student's t-tests on the raw data (or on log-transformed data depending on the degree and nature of skew in the data). Non-parametric alternatives, such as permutation tests, will be considered if the data are not approximately normal for any continuous outcome variables after log-transformation. A similar approach will be used for making pre vs. post treatment comparisons, when necessary, but with paired t-tests or their non-parametric alternatives. The response outcomes will be evaluated between treatment arms by Fisher's exact tests.

SECONDARY OUTCOMES:
Alterations in immunohistochemical (IHC) markers | Up to 6 months
  Pre- and post-treatment patient tumor samples will be compared. The study will compare data from patients treated with durvalumab and metformin to patients treated with Durvalumab alone and to patients from our own historical controls of head and neck squamous carcinoma (HNSCC), both untreated and treated with metformin monotherapy
Alterations in intratumoral immune cell populations | Up to 6 months
  The biomarker data will be compared for differences in means (or geometric means) between treatment arms using Student's t-tests on the raw data (or on log-transformed data depending on the degree and nature of skew in the data). Non-parametric alternatives, such as permutation tests, will be considered if the data are not approximately normal for any continuous outcome variables after log-transformation. A similar approach will be used for making pre vs. post treatment comparisons, when necessary, but with paired t-tests or their non-parametric alternatives.
Changes of the intratumoral immunophenotype and metabolism after exposure to durvalumab and metformin | Baseline up to 6 months
  The biomarker data will be compared for differences in means (or geometric means) between treatment arms using Student's t-tests on the raw data (or on log-transformed data depending on the degree and nature of skew in the data). Non-parametric alternatives, such as permutation tests, will be considered if the data are not approximately normal for any continuous outcome variables after log-transformation. A similar approach will be used for making pre vs. post treatment comparisons, when necessary, but with paired t-tests or their non-parametric alternatives.
Tumor size as measured by immune-related response criteria (irRC) | Up to 4 weeks post-treatment
  The biomarker data will be compared for differences in means (or geometric means) between treatment arms using Student's t-tests on the raw data (or on log-transformed data depending on the degree and nature of skew in the data). Non-parametric alternatives, such as permutation tests, will be considered if the data are not approximately normal for any continuous outcome variables after log-transformation. A similar approach will be used for making pre vs. post treatment comparisons, when necessary, but with paired t-tests or their non-parametric alternatives. The response outcomes will be evaluated between treatment arms by Fisher's exact tests.

OTHER OUTCOMES:
Assessment of alterations in metabolites produced in different tumor compartments | Up to 6 months
  The biomarker data will be compared for differences in means (or geometric means) between treatment arms using Student's t-tests on the raw data (or on log-transformed data depending on the degree and nature of skew in the data). Non-parametric alternatives, such as permutation tests, will be considered if the data are not approximately normal for any continuous outcome variables after log-transformation. A similar approach will be used for making pre vs. post treatment comparisons, when necessary, but with paired t-tests or their non-parametric alternatives.
Assessment of the interactions between the immune and metabolic microenvironments | Up to 6 months
  The biomarker data will be compared for differences in means (or geometric means) between treatment arms using Student's t-tests on the raw data (or on log-transformed data depending on the degree and nature of skew in the data). Non-parametric alternatives, such as permutation tests, will be considered if the data are not approximately normal for any continuous outcome variables after log-transformation. A similar approach will be used for making pre vs. post treatment comparisons, when necessary, but with paired t-tests or their non-parametric alternatives.
Circulating Tumor DNA | Baseline up to 12 days post surgery
  The possibility of measuring an increase in the release of circulating tumor DNA as an indicator of responsiveness or tumor progression is attractive and is supported by xenograft models. An attempt to correlate the mutations found in the circulating tumor DNA with the mutations in the tumor tissues will be performed. The identification of new mutations in circulating tumor DNA over time might inform the clinician about tumor evolution and provide evidence to support new treatment targets not identifiable in the primary tumor
Ultrasound and Photoacoustic Imaging | Baseline up to 38 days post visit 1.
  Our clinical project will evaluate diagnostic utility of multimodality imaging method of digital blood flow quantification based on 3D high frequency Doppler ultrasound and photoacoustic (PA) imaging in patients with Head and Neck Squamous cell carcinoma before and after treatment with Durvalumab and Metformin. This will be done to correlate changes in tissue and tumor oxygenation of the specific tumor of interest measured via photoacoustic imaging with treatment response.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Curry, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Curry J, Alnemri A, Philips R, Fiorella M, Sussman S, Stapp R, Solomides C, Harshyne L, South A, Luginbuhl A, Tuluc M, Martinez-Outschoorn U, Argiris A, Linnenbach A, Johnson J. CD8+ and FoxP3+ T-Cell Cellular Density and Spatial Distribution After Programmed Death-Ligand 1 Check Point Inhibition. Laryngoscope. 2023 Aug;133(8):1875-1884. doi: 10.1002/lary.30389. Epub 2022 Sep 20. PMID 36125263
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/